CLINICAL TRIAL: NCT06710509
Title: Patient Reminders Optimizing Mail-in Prevention Testing for Colorectal Cancer
Acronym: PROMPT-CRC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emily Rosenzweig (Industry)
Responsible Party: Sponsor-Investigator, Emily Rosenzweig, Director of Behavioral Science, Ascension Health
Organization: Ascension Health (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: RAS20240016
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Colon Cancer Screening
Keywords: colon cancer screening

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): Group not receiving the messages
- Experimental Group (Experimental): Group receiving the messages
  Interventions: Behavioral: Three Messaging Nudges

INTERVENTIONS:
Behavioral: Three Messaging Nudges — Patients in the Experimental Condition will receive a set of up to three email and text messages over the course of five days, while also receiving usual care which could include messaging from their practice or the electronic health record.
  Arms: Experimental Group

SUMMARY:
Screening is an important tool for early colorectal cancer detection, and the most recent evidence suggests that early detection significantly improves survival rates. Current medical guidelines recommend that all people aged 45 to 75 be screened regularly. However, actual rates of screening in the United States are much lower than this.

Colonoscopy is the gold standard in colon cancer screening, serving as both screening and prevention. However there are many barriers to colonoscopy uptake, including lack of awareness, patient reticence, scheduling complexity, and market variation in access. Stool testing is a valuable alternative to colonoscopy for low-risk patients. Exact Sciences is the company that makes Cologuard, which is the current best-in-class stool testing for colon cancer screening.

Despite being a convenient at-home screening option, patient engagement with screening via stool testing has room for improvement. Over 40% of Ascension patients who have a stool testing order placed for them never return the screening kit in the mail.

A large body of research demonstrates that interventions informed by behavioral science can support patients in engaging in a variety of preventative health behaviors. Personalized nudges have proven to be among the most effective types of interventions, along with interventions aimed at helping patients overcome barriers to screening. We aim to test whether behavioral nudges can increase stool testing kit return rates.

DETAILED DESCRIPTION:
Screening is an important tool for early colorectal cancer detection, and the most recent evidence suggests that early detection significantly improves survival rates. Current medical guidelines recommend that all people aged 45 to 75 be screened regularly. However, actual rates of screening in the United States are much lower than this, particularly among younger patient cohorts. Screening rates are still lower for patients who are "socially vulnerable" - a measure of the degree to which social and demographic factors make them vulnerable to health disparities.

Colonoscopy is the gold standard in colon cancer screening, serving as both screening and prevention. However there are many barriers to colonoscopy uptake, including lack of awareness, patient reticence, scheduling complexity, and market variation in access. Stool testing is a valuable alternative to colonoscopy for low-risk patients. Exact Sciences is the company that makes Cologuard, which is the current best-in-class stool testing for colon cancer screening.

Despite being a convenient at-home screening option, patient engagement with screening via stool testing has room for improvement. Over 40% of Ascension patients who have a stool testing order placed for them never return the screening kit in the mail.

A large body of research demonstrates that interventions informed by behavioral science can support patients in engaging in a variety of preventative health behaviors. Personalized nudges have proven to be among the most effective types of interventions, along with interventions aimed at helping patients overcome barriers to screening.4 We aim to test whether behavioral nudges can increase stool testing kit return rates.

ELIGIBILITY:
Inclusion Criteria:

* Age 45-75
* Have either a mobile phone number or an email address on file with the health system
* Included in and non-compliant on the Ascension Colon Cancer Screening Clinical Priority Goal measure.
* Have consented to receive electronic communications from the health system
* Ascension primary care provider placed an order for stool testing between 60 and 180 days prior to the intervention.
* No record of Cologuard stool testing lab results returned within 60 days of the order being placed.

Exclusion Criteria:

* Patients whose primary care providers are exempted from the campaign by the health system
* Patients with a record of having been screened for colorectal cancer through some other method during the time since the initial order for Cologuard stool testing was placed.
* Have received a nudge campaign from the Clinical Transformation team in the past 90 days
* Patients who have previously opted out of receiving electronic communications from the health system in our message delivery platform (Salesforce)

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2106 (Actual)
Dates: Start 2024-12-05 (Actual); Primary Completion 2025-01-02 (Actual); Study Completion 2025-02-26 (Actual)

PRIMARY OUTCOMES:
Percentage kit return at 4 weeks | 4 weeks from date first message was sent
  Percentage of patients who have Cologuard stool testing lab results returned 4 weeks after receiving the intervention

SECONDARY OUTCOMES:
Percentage kit return at 8 weeks | 8 weeks from date first message was sent
  Percentage of patients who have Cologuard stool testing lab results returned 8 weeks after receiving the intervention
Percentage kit return at 12 weeks | 12 weeks from date first message was sent
  Percentage of patients who have Cologuard stool testing lab results returned 12 weeks after receiving the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Emily Rosenzweig, Principal Investigator — Ascension Health
Locations (1):
- Ascension Health, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Has patient information that we are not approved to share